CLINICAL TRIAL: NCT07021651
Title: A Two-Center Randomized Controlled Trial
Brief Title: COMPARISON OF ERECTOR SPINA PLAN BLOCK AND THORACIC PARAVERTEBRAL BLOCK FOR PERIOPERATIVE ANALGESIA
Acronym: A Two-Center
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Anesthesiology and Reanimation Spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEM
Record Dates: First submitted 2025-06-04; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Paravertebral Block
MeSH Terms: interventions — Parapsychology

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erektor spina plan block (Active Comparator): The local anesthetic is injected into the fascial plane between the erector spinae muscle and the transverse processes of the vertebrae. This allows the anesthetic to spread cranially and caudally, affecting multiple spinal nerves
  Interventions: Procedure: Erector Spinae Plane (ESP) block admistring
- Toracik paravertebral block (Active Comparator): The local anesthetic is injected into the paravertebral space, which is bordered by the vertebral bodies, intervertebral discs, parietal pleura, and superior costotransverse ligament. This space contains the spinal nerves, sympathetic chain, and intercostal vessels
  Interventions: Procedure: Thoracic Paravertebral Block administring

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) block admistring — In the ESPB group, the probe was placed longitudinally at the level of the T5 transverse process, 2-3 cm lateral from the midline. The muscles were visualized superior to the transverse process ; then, the needle was inserted in the craniocaudal direction using the in-plane technique. A dose of 2 mL normal saline were injected into the two layers of the interfacial area under the erector spinae muscle, and the proper injection site was confirmed. After visualizing the linear spread of saline in the fascial plane, 20 mL of 0.25% bupivacaine was injected there for the block.
  Arms: Erektor spina plan block
Procedure: Thoracic Paravertebral Block administring — In the TPVB group, the probe was placed 2-3 cm laterally and vertically of the T5 spinous process. Once the transverse process, corresponding paravertebral space, internal intercostal membrane, and pleura was identified , the needle was inserted in the lateromedial direction using the in-plane technique. After confirmation of pleural displacement with 2 mL saline, 20 mL of 0.25% bupivacaine was administered for the block.
  Arms: Toracik paravertebral block

SUMMARY:
The primary aim of this study was to compare the postoperative analgesic efficacy of thoracic paravertebral block with erector spinae plane block, which we use in thoracotomy surgeries. Secondary aims were to compare these groups in terms of Riker Agitation-Sedation Scale (RASS) scores, postoperative complications, postoperative opioid consumption, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo thoracotomy and are between the ages of 18-65
* have American Society of Anesthesiologists (ASA) risk classification I-II will be included in the study.

Exclusion Criteria:

* Patients who did not agree to participate in the study,
* had an infection in the application area,
* had coagulopathy,
* were morbidly obese (Body mass index (BMI)>35),
* had drug allergy,
* had chronic pain, long-term opioid use, psychiatric illness history, and required emergency surgery were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Post-operative 30 minutes, 2 hours, 6 hours, 12 hours, 24 hours
  They will be numbered from 1 to 10. If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.

SECONDARY OUTCOMES:
Riker Agitation and Sedation Scale | Immediately after extubation
  7 Dangerous Agitation ... If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Patient satisfaction score: | Post-operative 30 minutes
  Patients' satisfaction with the quality of pain management will be assessed on the second postoperative day using the following scale: 1 = very dissatisfied; 2 = quite dissatisfied; 3 = moderate; 4 = quite satisfactory; 5 = very satisfactory.)
24-hour Tramadol usage: | posoperative 24 hours
  Amount of Tramadol used per 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Kayapınar, Di̇yarbakir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No